CLINICAL TRIAL: NCT06869603
Title: Evaluation of Adherence to the Mediterranean Diet in Patients with Recurrent Renal Stones and Disease Osteometabolic
Status: Recruiting | Type: Observational
Sponsor: IRCCS SYNLAB SDN (Other)
Collaborators: Department of Clinical Medicine and Surgery - University of Naples Federico II (Unknown)
Responsible Party: Sponsor
Other Study IDs: 3/23
Record Dates: First submitted 2024-03-25; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Renal Stones; Osteometabolic Disease
MeSH Terms: conditions — Nephrolithiasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The aim of this research protocol is to evaluate the adherence to the Mediterranean diet in patients suffering from recurrent kidney stones and osteometabolic diseases. Results of the study will allow to assess the dietary habits of patients with the above diseases. Given the universal prevalence of nephrolithiasis and osteometabolic diseases, the knowledge of these data appears crucial for the proper management of the dietary approach to prophylaxis secondar

ELIGIBILITY:
Inclusion Criteria:

* Patients with idiopathic relapsing nephrolithiasis with evidence instrumental of bilateral renal stones or emission of more than one stone in the past 5 years

Exclusion Criteria:

* Patients who had albumin-corrected plasma calcium levels > 11.0 mg/dl at the time of the first determination of serum levels of 25 OH vitamin D;
* Patients who had glomerular filtration rate < 60 mL/min/1.73 m2;
* Patients who had positive personal history of chronic granulomatous disease;
* pregnancy patients;
* Positive personal history for morphological abnormalities of the excretory system;
* incomplete data collection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with idiopathic relapsing nephrolithiasis with evidence instrumental of bilateral renal stones or emission of more than one stone in the past 5 years
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-12-07 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Patient eating habits | 1-36 months
  Questionaries to detect the patients eating habits.

CONTACTS AND LOCATIONS:
Locations (1):
- Irccs Synlab Sdn, Naples, Italy